CLINICAL TRIAL: NCT05400564
Title: Preventing Emotional and Behavioral Problems in Middle School Youth At-risk of Disability After the Covid-19 Pandemic With the Family Check-up Online
Brief Title: The Families and Middle School Success Project
Acronym: FMSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000404
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parenting; Parent-Child Relations; Self-regulation; Problem Behavior in School; School Adjustment; Depression
MeSH Terms: conditions — Self-Control; Depression

STUDY DESIGN:
Intervention Model Description: Families will be assigned to treatment vs. a school as usual control. The investigators will assess families at baseline and at 3-, 6-, 12- and 24- month follow ups. Families in the treatment condition will receive the intervention between baseline and the 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCU Online + Coach (Experimental): Parents in this arm will receive access to the FCU app and telehealth coaching/ support provided by a trained mental health provider. The FCU app includes a brief 5-minute assessment, feedback on parents' responses, and online tools to support parenting in areas that were identified as challenges by the assessment. These tools include videos, animated videos, parenting tips, and interactives to help practice parenting skills. Telehealth coaching sessions will focus on Healthy Behaviors, Positive Parenting, Rules and Consequences, School Support, and Communication.
  Interventions: Behavioral: Family Check-Up
- Control (No Intervention): Parents in this arm will receive school support as usual.

INTERVENTIONS:
Behavioral: Family Check-Up — This intervention includes access to the Family Check-Up app and telehealth coaching provided by trained mental health providers. Parents can contact their Coach as often as they like and a minimum of 3 coaching sessions will be scheduled.
  Arms: FCU Online + Coach

SUMMARY:
The purpose of the proposed research is to conduct an efficacy trial of the Family Check-Up (FCU) Online to prevent emotional and behavioral disorders among middle-school students at-risk for disability during the transition back to school after the COVID-19 pandemic. Mental health and behavior problems are at epidemic proportions as a result of the COVID-19 pandemic, with the highest rates in adolescents and children with disabilities. We propose to evaluate the efficacy of the FCU Online, a school-based, ecological approach to family intervention and risk reduction, across a group of students at-risk or identified with disability during the middle school years. The FCU Online for middle school youth has been evaluated in a randomized trial in prior research during the development of the program but has never been tested as a large-scale, school-based intervention or delivered by providers working in schools. It has recently been adapted for COVID-19 and includes new modules on coping with stress and home-to-school engagement to support the return to school after COVID-19 for students at-risk. Students in schools will be identified for services using indicators that are natural to the school environment (attendance, office discipline referrals, and grades), and will be followed for 2 years. We predict that engagement in the FCU Online will be associated with student reductions in emotional and behavior problems, improvements in academic skills, and improvements in attendance. Parenting skills such as home-to-school communication, positive parenting, and behavioral routines will be tested as mediators of intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A caregiver must have a child between the ages of 11 and 14
* The child must be a middle school student enrolled at a participating middle school including: Alder Creek Middle School in Milwaukee, Oregon, or Wilbur Rowe Middle School in Milwaukee, Oregon
* The caregiver must be the parent or legal guardian of the participating youth
* The caregiver must have a smartphone with text messaging capability and access to email
* The student must have one or more of the following risk factors: 1) two or more office discipline referrals; 2) grades below a 2.5 GPA; 3) poor attendance, i.e., missing more than 10% of school days; 4) IEP for emotional disturbance or related disabilities; or 5) concerns about the child on the behavioral and mental health screener (as indicated by a score of 3 on any one item, or a score of 2 or higher on at least two items).

Exclusion Criteria:

* The caregiver is unable to read in either English or Spanish
* The child is unable to complete the survey without parent's help
* The family is already participating in another study of the University of Oregon's Prevention Science Institute

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in family conflict (parent and child report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured with the CASEY
change from baseline in family relationships (parent and child report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured with the CASEY
change from baseline in child academic competence (parent, child and teacher report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured with the SSRS
change from baseline in child school engagement (parent, child and teacher report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured with the school participation measure
change from baseline in child's school grades (school report) | baseline, 3 months, 6 months, 12 months, 24 months
  Obtained via school records
change from baseline in child's achievement test scores/school records/IEP (school report) | baseline, 3 months, 6 months, 12 months, 24 months
  Obtained via school records
change from baseline in child's school attendance (school report) | baseline, 3 months, 6 months, 12 months, 24 months
  Obtained via school records
change from baseline in youth emotional problems (parent, child and teacher report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the SDQ
change from baseline in youth behavior problems (parent, child and teacher report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the SDQ
change from baseline in youth self regulation (parent, and child report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the SDQ
change from baseline in youth social/peer relationships (parent and child report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PASA
change from baseline in child's discipline referrals (school report) | baseline, 3 months, 6 months, 12 months, 24 months
  Obtained via school records

SECONDARY OUTCOMES:
change from baseline in parent depression and anxiety (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PHQ-9
change from baseline in parental stress (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PSS
change from baseline in youth depression (parent and child report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PHQ-9
change from baseline in parental sense of competency (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PSOC
change from baseline in positive parenting behaviors (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PCA
change from baseline in limit setting and supervision skills (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by the PCA
change from baseline in parenting involvement at school (parent report) | baseline, 3 months, 6 months, 12 months, 24 months
  Measured by a modified version of the home-based learning factor of the FIQ-EC

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stormshak, Ph.D., Principal Investigator — University of Oregon
Locations (1):
- University of Oregon Prevention Science Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the terms of the funding contract from IES, de-identified study data will eventually be deposited at a public repository, Inter-university Consortium for Political and Social Research (ICPSR), to increase its utility to qualified individuals within the scientific community. Direct requests for data from other researchers and the public will be also considered, and data will be made available in accordance with local institution policies, IRB recommendations, local/state/federal laws and regulations, and considerations for publication. Any applicable data sharing will follow HIPAA rules.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared at the end of the grant.
Access Criteria: In order to access these data, the ICPSR Data Archive will require a data use agreement (DUA), which will provide for (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. The data sharing agreement will also assure that the analysis being proposed is appropriate given the design and data available. This data will be shared with ICPSR and approved scientists without additional informed consent from the research participants.
URL: https://www.icpsr.umich.edu/

DOCUMENTS (1):
  • Informed Consent Form (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05400564/ICF_000.pdf